CLINICAL TRIAL: NCT05543525
Title: Advanced Myocardial Deformation Echocardiography for the Athlete's Heart Evaluation: Functional and Mechanistic Analysis
Brief Title: Myocardial Mechanics in Athlete's Heart
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); INSERM, CIC 1433 (Unknown)
Responsible Party: Principal Investigator, PACE Nathalie, Doctor of Medicine (MD) in Cardiology, Central Hospital, Nancy, France
Other Study IDs: 2022PI064
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Athlete Heart
Keywords: speckle tracking echocardiography; myocardial deformation; functional capacity; layer-specific strain
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male Athletes: Athletes who underwent a pre-participation medical evaluation in the Nancy University Hospital between January 1st, 2013, and January 1st, 2020.
  Interventions: Other: Echocardiography; Other: Cardiopulmonary exercise testing
- Control Group: A subgroup of 161 participants in a population-based cohort (STANISLAS Cohort) restricted by age and sex to create a control group in the current analysis.
  Interventions: Other: Echocardiography; Other: Cardiopulmonary exercise testing

INTERVENTIONS:
Other: Echocardiography — Transthoracic echocardiography
Other: Cardiopulmonary exercise testing — Cardiopulmonary exercise testing

SUMMARY:
Echocardiographic assessment of the endurance athletes' heart remains challenging due to a phenotypic overlap between reactive physiological adaptation and pathological remodelling. The lower range of normal values of lLeft ventricle systolic ejection fraction (LVEF) and global longitudinal strain (GLS) in athletes makes it difficult to differentiate changes related to adaptive remodelling or indicative of early cardiomyopathy.

This study aims to improve the assessment of athletes' hearts by identifying echocardiographic phenotypes, using a speckle tracking including temporal deformation pattern and layer-specific approach, and to define predictive factors of subtle LV systolic dysfunction and of mechanical LV abnormalities.

DETAILED DESCRIPTION:
Healthy male athletes belonging to local clubs, who underwent a pre-participation medical evaluation at the University Hospital of Nancy between 2013 and 2020, will be screened. Clinical, echocardiographic and cardiopulmonary exercise testing data will be compared to a group of healthy men from the STANISLAS cohort. Subtle LV dysfunction will be defined by a GLS <17.5%.

ELIGIBILITY:
Inclusion Criteria:

- athletes who underwent a pre-participation medical evaluation in the Nancy University Hospital between January 1st, 2013, and January 1st, 2020

Exclusion Criteria:

* female athletes,
* athletes followed for cardiomyopathy
* athletes who did not have transthoracic echocardiography (TTE) performed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cross-sectional study, using data from young high-performance athletes referred to the cardiologic department of Nancy University Hospital for a pre-participation medical evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Multilayer (= epi- and endocardial) left ventricular global longitudinal strain using Speckle-tracking echocardiography | Baseline
  expressed in %

SECONDARY OUTCOMES:
Age | Baseline
  years
Height | baseline
  meter
Weight | baseline
  meter
BMI | baseline
  kg/m²
Heart rate | baseline
  bpm
Type of practiced sport | baseline
  soccer, basketball, handball
Inter ventricular septum diameter | baseline
  mm
Left ventricle indexed mass | baseline
  g/m²
Left ventricular Ejection Fraction | baseline
  using simpson's biplane method, expressed in %
left ventricular End-diastolic volume | baseline
  ml
Cardiac Index | baseline
  ml/min/m²
Maximal E-wave velocity and Maximal A-wave velocity | baseline
  m/s
Left atrium End-systolic volume | baseline
  ml/m²
left ventricular global longitudinal strain (peak G) assessed by Speckle-tracking echocardiography | baseline
  expressed in %
PSI (pre stretch index) assessed by Speckle-tracking echocardiography | baseline
  expressed in %
PST (postsystolic thickening) assessed by Speckle-tracking echocardiography | baseline
  expressed in %
Peak VO2 | baseline
  L/min

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Pace, MD, Principal Investigator — CHRU Nancy
Locations (1):
- Chru Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.To achieve aims in the approved proposal. Proposals should be directed to n.pace@chru-nancy.fr.

REFERENCES:
- [Background] Spirito P, Pelliccia A, Proschan MA, Granata M, Spataro A, Bellone P, Caselli G, Biffi A, Vecchio C, Maron BJ. Morphology of the "athlete's heart" assessed by echocardiography in 947 elite athletes representing 27 sports. Am J Cardiol. 1994 Oct 15;74(8):802-6. doi: 10.1016/0002-9149(94)90439-1. PMID 7942554
- [Background] Caselli S, Maron MS, Urbano-Moral JA, Pandian NG, Maron BJ, Pelliccia A. Differentiating left ventricular hypertrophy in athletes from that in patients with hypertrophic cardiomyopathy. Am J Cardiol. 2014 Nov 1;114(9):1383-9. doi: 10.1016/j.amjcard.2014.07.070. Epub 2014 Aug 12. PMID 25217454
- [Background] Schnell F, Matelot D, Daudin M, Kervio G, Mabo P, Carre F, Donal E. Mechanical Dispersion by Strain Echocardiography: A Novel Tool to Diagnose Hypertrophic Cardiomyopathy in Athletes. J Am Soc Echocardiogr. 2017 Mar;30(3):251-261. doi: 10.1016/j.echo.2016.11.013. Epub 2017 Jan 5. PMID 28065584
- [Background] Abuli M, de la Garza MS, Sitges M. Differentiating Athlete's Heart from Left Ventricle Cardiomyopathies. J Cardiovasc Transl Res. 2020 Jun;13(3):265-273. doi: 10.1007/s12265-020-10021-8. Epub 2020 May 14. PMID 32410209
- [Background] Santoro A, Alvino F, Antonelli G, Caputo M, Padeletti M, Lisi M, Mondillo S. Endurance and Strength Athlete's Heart: Analysis of Myocardial Deformation by Speckle Tracking Echocardiography. J Cardiovasc Ultrasound. 2014 Dec;22(4):196-204. doi: 10.4250/jcu.2014.22.4.196. Epub 2014 Dec 26. PMID 25580194
- [Background] D'Ascenzi F, Solari M, Mazzolai M, Cameli M, Lisi M, Andrei V, Focardi M, Bonifazi M, Mondillo S. Two-dimensional and three-dimensional left ventricular deformation analysis: a study in competitive athletes. Int J Cardiovasc Imaging. 2016 Dec;32(12):1697-1705. doi: 10.1007/s10554-016-0961-6. Epub 2016 Aug 13. PMID 27522672
- [Background] Huttin O, Girerd N, Coiro S, Bozec E, Selton-Suty C, Lamiral Z, Frikha Z, Kobayashi M, Argulian E, Narula J, Fraser AG, Rossignol P, Zannad F. Association Between Layer-Specific Longitudinal Strain and Risk Factors of Heart Failure and Dyspnea: A Population-Based Study. J Am Soc Echocardiogr. 2019 Jul;32(7):854-865.e8. doi: 10.1016/j.echo.2019.03.011. Epub 2019 May 16. PMID 31104890